CLINICAL TRIAL: NCT05358002
Title: Comparative Study Between Frontalis Flap Advancement Versus Frontalis Sling Operations in Mangment of Congenital Blepharoptosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Hesham Ibrahim Abd ElFattah Ibrahim Shahin, Principal investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: MD-93-2020
Record Dates: First submitted 2022-04-09; First posted 2022-05-03 (Actual); Last update posted 2022-05-03 (Actual); Status verified 2022-04

CONDITIONS: Unrecognized Condition

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Frontalis sling (Active Comparator): Connecting the frontalis muscle action with the tarsus of the upper eyelid with synthetic material PTFE ( gore-tex )
  Interventions: Procedure: Frontalis flap
- Frontalis flap (Experimental): Fashonizing a flap from frontalis muscle and connecting it to the tarsus of the upper eyelid
  Interventions: Procedure: Frontalis flap

INTERVENTIONS:
Procedure: Frontalis flap — Fashonizing a flap from frontalis muscle and connecting it to the tarsus of the upper eyelid

SUMMARY:
A prospective comparative study between the results obtained by applying frontalis muscle flap advancement and frontalis sling operations for correction of congenital ptosis with poor levator muscle function. Study will include evaluation of the functional and cosmetic results, recurrence rates, and the incidence and varieties of different complications between the two techniques

DETAILED DESCRIPTION:
- Population of study & disease condition: Congenital ptosis with poor levator muscle function.

- Study setting: The ophthalmology unit of Abuelreesh Children Hospital.

- Inclusion criteria:

Criteria for inclusion in this study will be children more than 1 years age with:

1. moderate to severe ptosis with margin reflex distance1 (MRD1) ≤2 mm,
2. poor levator function of <4 mm,
3. good frontalis muscle function.

   * Exclusion criteria:

     1. Children with no Bell's phenomenon, the Marcus Gunn phenomenon, myasthenia gravis, strabismus, and blepharophimosis syndrome.
     2. Children with history of previous ptosis surgery or lid trauma.
   * Methodology in details:

Our study will be conducted on children with moderate to severe congenital ptosis with poor levator function attending the ophthalmology oculoplastic clinic of Abuelreesh children Hospital. At baseline, a detailed demographic and medical history will be collected, and the presence of an anomalous head posture is noted. All subjects will receive a complete preoperative ophthalmological evaluation. Slit-lamp examination, fundus examination and cycloplegic refraction will be done. Assessment of vision should be done according to the age, and the presence or absence of amblyopia is recorded. Best corrected visual acuity is also assessed if possible. Extraocular muscle functions will be evaluated for any associated abnormalities. All patients are tested for jaw winking syndrome and Bell's phenomenon.

The upper eyelid margin reflex distance (MRD1) will be measured which is the distance from the light reflex to the centre of the upper lid margin in primary position. The amount of ptosis is estimated by subtracting the MRD1 from 5 (5 - MRD1). The vertical interpalpebral fissure height will also be recorded. Measurement of levator muscle function is performed by measuring the excursion of the upper eyelid from downgaze to up gaze with the frontalis muscle fixed. Frontalis and orbicularis muscles functions are also assessed.

Patients will be divided randomly into two groups according to the technique used for correction of ptosis. We use the coin randomization method (Kang et al., 2008). Group A will undergo frontalis muscle flap advancement operation, while in group B, the children will be corrected by frontalis sling operation. Informed consent from the parents will be taken. All operations will be done under general anaesthesia and the incision sites will be marked using a surgical marker-pen in both techniques. Bupivacaine 0.5% with epinephrine 1:200,000 are infiltrated locally to improve intraoperative haemostasis and postoperative analgesia.

Surgical steps of frontalis muscle flap advancement technique:

1. A lid-crease incision is made 4-5 mm above the lash line or according to the height of the opposite lid crease starting lateral to the supraorbital notch.
2. The incision is made deep to the plane beneath the orbicularis oculi and the dissection is upward as far as 0.5-1 mm above the superior margin of the eyebrow.
3. A strip of orbicularis, about 1-2 mm wide, is excised from the lower margin of the incision exposing the anterior surface of the tarsal plate.
4. Two parallel cuts, 1.5-2 cm apart, are made cephalad at the middle third of the myofascial tissue between the two dissected planes, forming a superiorly based rectangular myofascial flap that can be drawn downward freely.
5. A 15×20mm quadrangular frontalis muscle flap is dissected and pulled down. The free flap border is then attached to the upper third of tarsal plate with three 6-0 polypropylene sutures.
6. The central suture (highest point) determines the level of the upper-eyelid margin (just nasal to the pupil level). The eyelid margin is set at or 1 mm above the limbus.
7. The medial and lateral sutures are attached at the level of the medial and lateral limbus, respectively. Two additional sutures are applied along the line of fixation to form a smooth line if necessary.
8. After adjusting the fixation level properly, the redundant muscle is trimmed and the skin is closed with polypropylene 6-0 continuous suture.
9. A compressive patch will be applied for 24 hours.

Surgical steps of frontalis sling operation:

1. An eyelid spatula with ointment will be placed under the ptosed lid to prevent ocular trauma during skin incision and when the needle is passed.
2. Three stab incisions (3mm) in the lid will be made 2 mm from the lid margin. These incisions will be done through the skin and orbicularis muscle to expose the tarsus.
3. Two brow incisions, down to the level of periosteum, will be made just above the brow hairs, approximately in line with the lateral and medial canthi.
4. A forehead incision approximately (8-10 mm) above the brow, down to periosteum, will be placed midway between the 2 brow incisions.
5. A pocket will be dissected superiorly beneath the frontalis muscle, with blunt scissors, in the central forehead incision.
6. Sling material stringing will be performed using Wright needle.
7. Frontalis sling suspension will be done using Crawford procedure (double triangle configurations).
8. The sling material used will be polytetrafluoroethylene (PTFE) 2-0 suture material.
9. The lid contour and height will be adjusted by pulling on the ends of sling material. The eyelid margin is elevated to (or 1 mm above) the superior limbus of the cornea. The nasal third will be slightly higher than the lateral third.
10. Both ends of the sling will be tied together. The ends of sling material will be trimmed about 3 mm from the knot and the knot is buried into the preformed pocket.
11. The brow and forehead skin incisions are closed using 6-0 polyglycolic 610 sutures. In both groups, All patients will be prescribed topical antibiotic ointment for skin wounds for one week. Frequent lubricant eye drops every 1 hour and lubricant gel every 2 hours and before sleeping, will be applied for the early postoperative period. Then the medication intervals will be adjusted according to lagophthalmos and exposure keratopathy. The sutures will be removed 5-7 days after surgery. In group A, after the third day, alternating eyelid opening (with the frontalis muscle) and closing movements (with the orbicularis muscle) are started to reduce adherence of the muscle flap to the surrounding structures.

Patients will be seen for follow-up at the second postoperative day, 1 month, 3 months and 6 months. Our follow up will include MRD1, amount of residual ptosis, lid contour, cycloplegic refraction, lagophthalmos and corneal exposure, state of the scar, asymmetry of lid position in unilateral cases and other complications

ELIGIBILITY:
Inclusion Criteria:

* cases of congenital ptosis

Exclusion Criteria:

* associated with other anomalies e.g: blepharophimosis syndrome , marcus gunn jaw winking.
* previous ptosis surgery.

Ages: 1 Year to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 40 (Actual)
Dates: Start 2020-05-20 (Actual); Primary Completion 2022-04-09 (Actual); Study Completion 2022-04-09 (Actual)

PRIMARY OUTCOMES:
Improvement of MRD ( marginal reflex distance ) | About 6 months
  Improvement of the marginal reflex distance that is measured by the ruler, which is the distance between the margin of the upper eyelid and the light reflex reflecting from the cornea from a torch against the cornea

SECONDARY OUTCOMES:
Improvement of the vertical palpebral fissure height | 6 months
  Measuring the distance between margin of the upper and lower eyelid using a ruler

CONTACTS AND LOCATIONS:
Overall Officials: Magda S Abdelaziz, Prof., Principal Investigator — Kasr alainy
Locations (1):
- Kasr al ainy, Cairo, Egypt